CLINICAL TRIAL: NCT02099591
Title: A Phase I, Open-Label, Multicentre Study to Assess the Pharmacokinetics and Safety of Naloxegol in Paediatric Patients Ages ≥ 6 Months to < 18 Years Receiving Treatment With Opioids
Brief Title: Phase I Pharmacokinetics and Safety Study of Naloxegol in Paediatric OIC Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kyowa Kirin Pharmaceutical Development Ltd (Industry)
Responsible Party: Sponsor
Organization: Kyowa Kirin Co., Ltd. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D3820C00016; UTN: U1111-1154-5575 (Other: World Health Organization); 2013-003935-32 (EudraCT Number)
Record Dates: First submitted 2014-02-13; First posted 2014-03-31 (Estimated); Last update posted 2024-06-17 (Actual); Status verified 2024-06

CONDITIONS: Constipation, Signs and Symptoms, Digestive
Keywords: Constipation; Colonic Inertia; Dyschezia; Pharmacokinetics; Naloxegol; Paediatric; Opioids; Opioid induced constipation; OIC; Phase 1
MeSH Terms: conditions — Constipation; Opioid-Induced Constipation | interventions — naloxegol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- Age group: > = 12y to < 18y - Lower dose (Experimental): Naloxegol Dose equivalent to 12.5mg in adults which will be administered once daily for up to 6 months.
  Interventions: Drug: Naloxegol
- Age group: > = 12y to < 18y - Higher dose (Experimental): Naloxegol Dose equivalent to 25mg in adults which will be administered once daily for up to 6 months.
  Interventions: Drug: Naloxegol
- Age group: > = 6y to < 12y - Lower dose (Experimental): Naloxegol Dose equivalent to 12.5mg in adults which will be administered once daily for up to 6 months.
  Interventions: Drug: Naloxegol
- Age group: > = 6y to < 12y - Higher dose (Experimental): Naloxegol Dose equivalent to 25mg in adults which will be administered once daily for up to 6 months.
  Interventions: Drug: Naloxegol
- Age group: > = 6mo to < 6y - Lower dose (Experimental): Naloxegol Dose equivalent to 12.5mg in adults which will be administered once daily for up to 6 months.
  Interventions: Drug: Naloxegol
- Age group: > = 6mo to < 6y - Higher dose (Experimental): Naloxegol Dose equivalent to 25mg in adults which will be administered once daily for up to 6 months.
  Interventions: Drug: Naloxegol

INTERVENTIONS:
Drug: Naloxegol — Opioid Antagonist
  Other Names: Moventig

SUMMARY:
To characterize the pharmacokinetics (PK) of naloxegol after single oral dose and through population PK in paediatric patients with opioid induced constipation (OIC) or at risk of OIC.

ELIGIBILITY:
Main inclusion criteria, patient with:

* malignant or non-malignant pain who are receiving or (are about to receive) acute or chronic treatment with opioids
* newly diagnosed constatipation, with history of constipation treated with laxatives or expected to develop constipation after opioid treatment
* ability to be present in the clinic for at least 10 hours following the first study drug for blood sampling and to return at 24 hours for blood sampling.

Main exclusion criteria:

* Current acute or chronic use of methadone
* History of an neoplasm or an ongoing gastrointestinal-related issue
* Signs or symptoms of gastrointestinal obstruction
* History of prolonged neutropenia or thrombocytopenia with clinical sequelae.
* Patients currently receiving the first cycle of chemotherapy

Ages: 6 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 61 (Actual)
Dates: Start 2014-11 (Actual); Primary Completion 2021-04 (Actual); Study Completion 2021-04 (Actual)

PRIMARY OUTCOMES:
To characterise the pharmacokinetics of naloxegol after single oral dose and through population pharmacokinetics in paediatric patients with opioid induced constipation | Day 1 : Pre-dose (within 30 min prior to drug dosing), 0.5, 1, 2, 4, 6, 8, 10 and 24 hours

SECONDARY OUTCOMES:
To characterise the pharmacokinetics of naloxegol after multiple, once-daily, oral dosing in paediatric opioid induced constipation patients who continue participation beyond Day 1 | Day 7 (minimum 3 days of naloxegol treatment): pre-dose and 4 hours post-dose
Palatability of naloxegol liquid drug formulation | Day 1 and Day 2 after dose
Ability of the patient to swallow the tablet | Day 1 and Day 2 after dose
Clinical outcome measures by assessment of laxative use | From Day 1 until the End of treatment (26 week of study)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Davies, Principal Investigator — Nottingham Children's Hospital
Locations (16):
- Odense University Hospital, Odense, Denmark
- Israel (2):
  - Rambam Medical Center, Oncology Institute, Haifa
  - Schneider Children Medical Center, Petah Tikva
- Norway (3):
  - Haukeland Universitetssykehus, Bergen
  - Oslo University Hospital - Rikshospitalet, Oslo
  - St. Olavs Hospital, Trondheim
- Spain (5):
  - Pediatric Oncology Unit Hospital Vall d'Hebron, Barcelona
  - Hospital Infantil Universitario Nino Jesus, Madrid
  - Hospital Universitario Madrid Sanchinarro, Madrid
  - Unidad de Hematología y Oncología Pediátrica - Hospital Universitario HM Monteprincipe, Madrid
  - Hospital Universitario Virgen de la Arrixaca, Murcia
- United Kingdom (5):
  - The Leeds Teaching Hosptial NHS Trust, Leeds
  - Alder Hey Children's Hospital, Liverpool
  - Royal Marsden Hospital, London
  - Nottingham Children's Hospital, Nottingham
  - Oxford University Hospitals NHS Foundation Trust, Oxford